CLINICAL TRIAL: NCT03432897
Title: BrUOG 337: Olaparib Prior to Radical Prostatectomy For Patients With Locally Advanced Prostate Cancer and Defects in DNA Repair Genes
Brief Title: BrUOG 337: Olaparib Prior to Radical Prostatectomy For Advanced Prostate Cancer Defects in DNA Repair Genes
Acronym: 337
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment secondary to eligibility criteria
Sponsor: Brown University (Other)
Collaborators: Rhode Island Hospital (Other); The Miriam Hospital (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 337
Record Dates: First submitted 2017-10-05; First posted 2018-02-14 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate
Keywords: High risk; Defects; prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Olaparib 300 mg BID q 4 weeks for up to 3 cycles. The 3rd cycle will not be given if patient is found to progress post cycle 2.
  Between 22-42 days post Olaparib, patients will undergo a prostatectomy.
  Interventions: Drug: Olaparib Pill; Procedure: Prostatectomy

INTERVENTIONS:
Drug: Olaparib Pill — 300 mg BID
Procedure: Prostatectomy — 22-42 days post Olaparib patients will undergo surgery

SUMMARY:
This study will evaluate approximately 3 months of treatment with the drug olaparib in patients with prostate cancer. A capsule formulation of olaparib (tradename Lynparza™) is approved by the United States Food and Drug Administration (FDA) for the treatment of women with advanced BRCA-mutated ovarian cancer. Olaparib is an investigational drug in prostate cancer. A tablet formulation of olaparib is being tested in this study. It is a new formulation which is more convenient for patients than the approved capsule formulation because fewer tablets of olaparib need to be taken daily than with capsules.

The purpose of the study is to evaluate whether olaparib can reduce prostate cancer with defects in DNA repair genes when olaparib is given for approximately 3 months before surgery.

DETAILED DESCRIPTION:
1.1 Primary Objective 1.1.1. To evaluate the Prostate Specific Antigen (PSA) response rate of olaparib prior to radical prostatectomy for patients with locally advanced prostate cancer and defects in DNA repair genes.

1.2 Secondary Objectives 1.2.1 To evaluate the PSA progression-free survival of olaparib and radical prostatectomy for patients with locally advanced prostate cancer and defects in DNA repair genes.

1.2.2 To evaluate the safety of olaparib prior to radical prostatectomy for patients with locally advanced prostate cancer

1.2.3 To evaluate the rate of defects in DNA repair genes in patients with newly diagnosed locally advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed adenocarcinoma of the prostate.
* High risk for recurrence after prostatectomy including any of the following

  * Lymph node involvement by radiographic criteria
  * T3 or T4 disease by radiographic criteria
  * T2 disease and either PSA > 20 or Gleason 8,9 or 10
* Defects in any of the following genes:BRCA1, BRCA 2, ATM, CHEK1, CHEK2, FANCONIS ANEMIA (FANCL), HDAC2, PALB2, BARD1, BRIP1, CDK12, PPP2R2A, RAD51B, RAD51C, RAD51D, or RAD54L as assessed by Foundation Medicine FoundationOne assay on tumor tissue or cell-free DNA from peripheral blood via the FoundationACT assay.
* No distant visceral metastases.
* No prior chemotherapy or radiation for prostate cancer or PARP inhibitor. Prior and current hormone therapy (< 6 months from start date on study) for prostate cancer is allowed. Patients are allowed to remain on hormone therapy on study.
* ECOG performance status 0-1.
* Age>18.
* Required entry laboratory parameters

  * ANC≥ 1,500 cells/mm3;
  * Hemoglobin > 10.0g/dL with no blood transfusion in the last 14 days
  * Platelet count ≥100 x 109/L,
  * Total bilirubin ≤ 1.5 x ULN,
  * AST and ALT ≤ 2.5 x ULN
  * Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min
* Life expectancy of at least 1 year as documented by treating physician.
* All Men must be willing to consent to using two highly effective contraception while on treatment and for at least 4 months (120 days) after last treatment on study
* Signed study-specific consent form prior to study entry.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations- to be documented and submitted to BrUOG.
* Formalin fixed, paraffin embedded (FFPE) tumor sample from the primary cancer must be available for central testing coordinated by Rhode Island Hospital pathology. If there is not written confirmation of the availability of an archived tumor sample prior to enrollment the patient is not eligible for the study. Submit this written certification to BrUOG
* Patient agreed to not receiving any live virus and live bacterial vaccines while receiving study medication and during the 30 day follow up period. Patient should be made aware of this and it should be documented to BrUOG.
* Patient agreed to not consume grapefruit juice while on study treatment. Submit documentation patient was instructed and agreed.

Exclusion Criteria:

* Participation in another clinical study with an investigational anticancer product during the last 2 months (from day 1 of treatment on this trial). This pertains to treatment no trials the patient may only be seen in follow-up.
* Any previous treatment with PARP inhibitor for this or another cancer, including olaparib.
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer or other solid tumors including lymphomas (without bone marrow involvement) which was curatively treated with no evidence of disease for ≥5 years. Diagnosis date and treatment confirmation required to be sent to BrUOG. Certification from treating physician that patient is disease free is required.
* Resting ECG with QTc > 470 msec on 2 time-points within a 24 hour period or known family history of long QT syndrome
* Patients receiving any systemic chemotherapy or radiotherapy within 3 weeks prior to study treatment
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Concomitant use of the substrates of CYP3A4, CYP1A2, 2B6, 2C9, 2C19 and P-gp should be cautioned while on study.

CYP3A4 - hormonal contraceptive, simvastatin, cisapride, cyclosporine, ergot alkaloids, fentanyl, pimozide, sirolimus, tacrolimus and quetiapine CYP1A2 - duloxetine, melatonin CYP2B6 - bupropion, efavirenz CYP2C9 - warfarin CYP2C19 - lansoprazole, omeprazole, S-mephenytoin P-gp - simvastatin, pravastatin, digoxin, dabigatran, colchicine OATP1B1 - bosentan, glibenclamide, repaglinide, statins and valsartan OCT1, MATE1, MATE2K - metformin OCT2 - serum creatinine OAT3 -furosemide, methotrexate

* Persistent toxicities deemed related to previous cancer therapy, excluding alopecia.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with brain metastases.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any prior major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Immunocompromised patients that according to treating investigator would increase their risk to protocol treatment, or Patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable as long as not within 28 days from study registration).
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for prostate cancer, therefore male participants only, are allowed.
Enrollment: 1 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mega, MD, Principal Investigator — BrUOG
Locations (1):
- Lifespan Cancer Institute: The Miriam and Rhode Island Hospitals, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nientiedt C, Duensing A, Zschabitz S, Jager D, Hohenfellner M, Stenzinger A, Duensing S. PARP inhibition in prostate cancer. Genes Chromosomes Cancer. 2021 May;60(5):344-351. doi: 10.1002/gcc.22903. Epub 2020 Oct 28. PMID 33084183

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Olaparib 300 mg BID q 4 weeks for up to 3 cycles. The 3rd cycle will not be given if patient is found to progress post cycle 2.
  Between 22-42 days post Olaparib, patients will undergo a prostatectomy.
  Olaparib Pill: 300 mg BID
  Prostatectomy: 22-42 days post Olaparib patients will undergo surgery
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Prostate Specific Antigen (PSA) Response
Description: Response:Reduction of at least 50% in the prostate-specific antigen level from baseline Progression:A 25% increase in PSA from baseline
  Baseline then approximately 8 weeks later and 2 weeks post Olaparib, approximately 10-14 weeks after baseline and then approximately every 6 months for 2 years in follow-up.
Time Frame: Throughout the trial for approximately 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: PSA Progression-free Survival of Olaparib and Radical Prostatectomy for Patients With Locally Advanced Prostate Cancer and Defects in DNA Repair Genes.
Description: Evaluation by treating physician
Time Frame: Post treatment (approximately 8-12 weeks) and approximately every 6 months for 2 years.
Measure: Number; unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 1
months | 7

3. Secondary Outcome: Safety of Olaparib Prior to Radical Prostatectomy for Patients With Locally Advanced Prostate Cancer
Time Frame: Eight to 12 weeks prior to radical prostatectomy utilizing the descriptions and grading scales found in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 for grading all adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: From time of informed consent and until 4 weeks (30 days (+7 days)) after the patient has stopped study participation/treatment (olaparib or surgery, whatever is the last date of treatment), maximum of 20 weeks.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=1)
Dysgeusia (Nervous system disorders) | 1
Bronchial infection (Infections and infestations) | 1
Localized edema (General disorders) | 1
Edema limbs (General disorders) | 1
Malaise (General disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Fatigue (General disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03432897/Prot_SAP_ICF_000.pdf